CLINICAL TRIAL: NCT00304915
Title: HIV Translating Initiatives for Depression Into Effective Solutions
Acronym: HI-TIDES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNT 05-152
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: HIV, Depression
Keywords: HIV, depression; patient care management; patient care team
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Collaborative Care Intervention (Experimental): HIV patients were screened for depression and the screener results were available to HIV clinicians. Depressed HIV patients received collaborative care intervention.
  Interventions: Behavioral: Collaborative Care Interventions
- Arm 2: Usual Care (No Intervention): HIV patients were screened for depression and the screener results were available to HIV clinicians. Depressed HIV patients received usual care.

INTERVENTIONS:
Behavioral: Collaborative Care Interventions — Patients in the intervention group will be supported by a depression collaborative care team that will include a depression nurse care manager, clinical pharmacist, and psychiatrist. The depression nurse care manager will evaluate depression symptom severity, antidepressant side effects, depression and HIV medication adherence every two weeks over the phone during the acute phase of treatment and will record these results in CPRS. After a 50% improvement in depression severity, the intervention subject will move into the continuation phase of treatment and the patient will be contacted every four weeks by the depression nurse case manager.
  Arms: Arm 1: Collaborative Care Intervention

SUMMARY:
This study is a randomized trial designed to test and refine a collaborative care model for treating depression in VA patients with HIV.

DETAILED DESCRIPTION:
Background: Depression is the most common mental disorder in HIV infected patients. Despite the availability of efficacious treatments for depression, evidence suggests that it is under-diagnosed and under-treated in routine HIV care. To address this problem, the investigators will adapt and implement a collaborative stepped-care model for depression treatment in HIV clinics. This proposal builds on past success of the TIDES/WAVES programs used in VA primary care. The project (HI-TIDES or HIV Translating Initiatives for Depression into Effective Solutions) will implement the primary care collaborative care model for depression treatment in HIV clinics using evidence-based implementation strategies. Objectives: The objectives of this proposal are to: 1) Develop and evaluate the process of adapting, implementing, and sustaining collaborative care for depression in VA HIV clinics, 2) Compare the quality of depression care and the clinical effectiveness of HI-TIDES to usual care in the HIV clinics, and 3) Evaluate the cost-effectiveness of patients assigned to HI-TIDES relative to patients assigned to usual care in HIV clinics. Methods: The implementation framework for this proposal is primarily informed by the Rogers diffusion of innovation model, Simpson Transfer Model, and the PRECEDE model. The VA and American Psychiatric Association Practice Guidelines inform the stepped care collaborative model intervention as source documents for summarizing the evidence for depression treatment for the general population. An expert panel will be convened to rate the quality of available evidence for depression treatment in the context of HIV. Patients will be recruited from VA HIV clinics: Little Rock, Atlanta, and Houston. The intervention will be randomized at the level of the patient. The investigators expect to recruit a total of 140 intervention and 140 usual care patients. Patients in the intervention group will be supported by a depression collaborative care team that will include a depression nurse care manager, clinical pharmacist, and psychiatrist. The depression nurse care manager will evaluate depression symptom severity, antidepressant side effects, depression and HIV medication adherence every two weeks over the phone during the acute phase of treatment and will record these results in the VA electronic medical record. After a 50% improvement in depression severity, the intervention subject will move into the continuation phase of treatment and the patient will be contacted every four weeks by the depression nurse case manager. A formative evaluation will occur during start-up and throughout the implementation of the intervention. A summative evaluation will document the effectiveness and cost-effectiveness of the intervention using an intent to treat analysis plan. Findings: No results at this time. Status: Start-up activities. Impact: The proposed study is highly relevant to the VA and the Veterans it serves for many reasons. First, the majority of VA patients with HIV are not seen in the primary care clinics and therefore will not benefit from VA's efforts in primary care settings to improve depression identification and treatment. Second, in addition to the negative outcomes of depression generally, depression in HIV patients is associated with additional negative outcomes including accelerated HIV disease progression, decreased immune system functioning, and premature death. Third, directly moving collaborative depression care from primary care clinics to HIV clinics is likely to fail for several reasons including the comorbidities associated with depressed HIV patient and the potential for drug-drug interactions. The proposed project will address these gaps and provide effectiveness and cost-effectiveness analyses to inform decisions about larger scale implementation of the HI-TIDES intervention.

ELIGIBILITY:
Inclusion Criteria:

1. current 9-item Patient Health Questionnaire (PHQ-9) score of 10 or more and
2. current treatment in the HIV clinic.

Exclusion Criteria:

1. patients who do not have access to a telephone,
2. patients with current suicidal ideation,
3. patients with significant cognitive impairment as indicated by a score < 10 on the HIV Dementia Scale, and
4. patients with a chart diagnosis of schizophrenia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2007-02; Primary Completion 2009-07 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Pyne, MD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (3):
- United States (3):
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Arkansas
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Investigators can request IPD by contacting the PI.

REFERENCES:
- [Result] Pyne JM, Asch SM, Lincourt K, Kilbourne AM, Bowman C, Atkinson H, Gifford A. Quality indicators for depression care in HIV patients. AIDS Care. 2008 Oct;20(9):1075-83. doi: 10.1080/09540120701796884. PMID 18825515
- [Result] Fortney JC, Pyne JM, Smith JL, Curran GM, Otero JM, Enderle MA, McDougall S. Steps for implementing collaborative care programs for depression. Popul Health Manag. 2009 Apr;12(2):69-79. doi: 10.1089/pop.2008.0023. PMID 19320606
- [Result] Ackerman B, Pyne JM, Fortney JC. Challenges associated with being an off-site depression care manager. J Psychosoc Nurs Ment Health Serv. 2009 Apr;47(4):43-9. doi: 10.3928/02793695-20090401-01. PMID 19437931
- [Result] Pyne JM, Fortney JC, Curran GM, Tripathi S, Atkinson JH, Kilbourne AM, Hagedorn HJ, Rimland D, Rodriguez-Barradas MC, Monson T, Bottonari KA, Asch SM, Gifford AL. Effectiveness of collaborative care for depression in human immunodeficiency virus clinics. Arch Intern Med. 2011 Jan 10;171(1):23-31. doi: 10.1001/archinternmed.2010.395. PMID 21220657
- [Result] Curran GM, Pyne J, Fortney JC, Gifford A, Asch SM, Rimland D, Rodriguez-Barradas M, Monson TP, Kilbourne AM, Hagedorn H, Atkinson JH. Development and implementation of collaborative care for depression in HIV clinics. AIDS Care. 2011 Dec;23(12):1626-36. doi: 10.1080/09540121.2011.579943. Epub 2011 Jun 30. PMID 21714689
- [Result] Fortney JC, Pyne JM, Steven CA, Williams JS, Hedrick RG, Lunsford AK, Raney WN, Ackerman BA, Ducker LO, Bonner LM, Smith JL. A Web-based clinical decision support system for depression care management. Am J Manag Care. 2010 Nov;16(11):849-54. PMID 21348556
- [Result] Chapman J, Oser M, Hockemeyer J, Weitlauf J, Jones S, Cheung R. Changes in depressive symptoms and impact on treatment course among hepatitis C patients undergoing interferon-alpha and ribavirin therapy: a prospective evaluation. Am J Gastroenterol. 2011 Dec;106(12):2123-32. doi: 10.1038/ajg.2011.252. Epub 2011 Aug 9. PMID 21826113
- [Result] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Result] Bottonari KA, Tripathi SP, Fortney JC, Curran G, Rimland D, Rodriguez-Barradas M, Gifford AL, Pyne JM. Correlates of antiretroviral and antidepressant adherence among depressed HIV-infected patients. AIDS Patient Care STDS. 2012 May;26(5):265-73. doi: 10.1089/apc.2011.0218. Epub 2012 Mar 21. PMID 22536930
- [Result] Painter JT, Fortney JC, Gifford AL, Rimland D, Monson T, Rodriguez-Barradas MC, Pyne JM. Cost-Effectiveness of Collaborative Care for Depression in HIV Clinics. J Acquir Immune Defic Syndr. 2015 Dec 1;70(4):377-85. doi: 10.1097/QAI.0000000000000732. PMID 26102447
- See also: PubMed — http://www.ncbi.nlm.nih.gov/pubmed/26126749

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Collaborative Care Intervention: Collaborative Care Intervention: Patients in the intervention group will be supported by a depression collaborative care team that will include a depression nurse care manager, clinical pharmacist, and psychiatrist. The depression nurse care manager will evaluate depression symptom severity, antidepressant side effects, depression and HIV medication adherence every two weeks over the phone during the acute phase of treatment and will record these results in VA electronic medical record. After a 50% improvement in depression severity, the intervention subject will move into the continuation phase of treatment and the patient will be contacted every four weeks by the depression nurse case manager.
- Arm 2: Usual Care: Usual care arm. Usual care will include depression screening with the same 9-item Patient Health Questionnaire (PHQ-9) screener used for Arm 1. The HI-TIDES depression care team will not be a part of the usual care condition.
Period: Overall Study
Arm/Group | Arm 1: Collaborative Care Intervention | Arm 2: Usual Care
Started | 123 | 126
Completed | 105 | 110
Not Completed | 18 | 16
Not completed — Lost to Follow-up | 11 | 11
Not completed — Death | 4 | 5
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Collaborative Care Intervention: Collaborative Care Intervention: Patients in the intervention group will be supported by a depression collaborative care team that will include a depression nurse care manager, clinical pharmacist, and psychiatrist. The depression nurse care manager will evaluate depression symptom severity, antidepressant side effects, depression and HIV medication adherence every two weeks over the phone during the acute phase of treatment and will record these results in CPRS. After a 50% improvement in depression severity, the intervention subject will move into the continuation phase of treatment and the patient will be contacted every four weeks by the depression nurse case manager.
- Arm 2: Usual Care: Usual care arm. Usual care will include depression screening with the same PHQ-9 screener used for Arm 1. The HI-TIDES depression care team will not be a part of the usual care condition.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Collaborative Care Intervention | Arm 2: Usual Care | Total
Number analyzed (Participants) | 123 | 126 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (8.7) | 49.8 (10.5) | 49.8 (9.6)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 120 | 122 | 242
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 78 | 77 | 155
  White | 45 | 49 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Depression Treatment Response
Description: Depression symptom severity over the past two weeks was measured using the Hopkins Symptom Checklist (SCL-20). The SCL-20 includes the 13-item depression scale plus 7 depression-related items from the Hopkins Symptom Checklist-90-Revised. The items are scored from 0 to 4 and averaged to provide a mean depression severity score from 0 to 4. Depression treatment response at 6-months was defined as a 50% decrease in mean SCL-20 score compared to baseline.
Time Frame: 6 months
Population: intent to treat analysis
Measure: Number; unit: percent response
Arm/Group | Arm 1: Collaborative Care Intervention | Arm 2: Usual Care
Number analyzed (Participants) | 123 | 126
percent response | 33.3 | 17.5
Statistical Analysis 1: Comparison: Arm 1: Collaborative Care Intervention vs Arm 2: Usual Care; Test type: Superiority or Other; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 2.5, 95% CI 2-sided [1.37 to 4.56]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm 1: Collaborative Care Intervention | Arm 2: Usual Care
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/126
Other Adverse Events (participants affected / at risk) | 0/123 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes